CLINICAL TRIAL: NCT01798914
Title: Patient Transfer Program for Transitioning From Exubera® (Insulin Human [rDNA Origin]) Inhalation Powder to Technosphere® Insulin (Insulin Human [rDNA Origin]) Inhalation Powder
Brief Title: Patient Transitioning From Exubera® Inhalation Powder to Technosphere® Insulin Inhalation Powder
Status: No longer available | Type: Expanded Access
Sponsor: Mannkind Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: MKC-TI-139
Record Dates: First submitted 2013-02-19; First posted 2013-02-26 (Estimated); Last update posted 2016-01-20 (Estimated); Status verified 2016-01

CONDITIONS: Type 1 Diabetes; Type 2 Diabetes
MeSH Terms: conditions — Diabetes Mellitus, Type 1; Diabetes Mellitus, Type 2

INTERVENTIONS:
Drug: Technosphere Insulin Inhalation Powder — Patient Transitioning From Exubera® Inhalation Powder to Technosphere® Insulin Inhalation Powder
  Other Names: Afrezza Inhalation Powder

SUMMARY:
The purpose of this study is to allow patients with specific needs for inhaled insulin to continue with inhaled insulin therapy using Technosphere Insulin after Exubera was withdrawn from the market.

DETAILED DESCRIPTION:
A Phase 3, open label, multicenter, safety follow up trial to convert the treatment of subjects currently using Exubera to treatment with TI Inhalation Powder

ELIGIBILITY:
Inclusion Criteria:

* Subject has type 1 or type 2 diabetes mellitus and is currently being treated with or has been treated with Exubera.
* Subject has a severe phobia to sc injections of insulin (needle phobia) preventing conventional treatment OR has impaired sc insulin absorption

Exclusion Criteria:

* Smoking in the previous 6 months
* History of asthma or chronic obstructive pulmonary disease (COPD) or any other significant pulmonary disease, or exposure to pulmonary toxins.
* Clinically significant pulmonary abnormalities on chest high-resolution computed tomography (HRCT).
* PFT results prior to transferring to TI Inhalation Powder showing any of the following: FEV1 < 70% of predicted, FVC < 70% of predicted, DLCO < 70% of predicted, TLC < 80% of predicted.
* Allergy to insulin

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Dates: Start 2008-10; Primary Completion 2015-04 (Actual); Study Completion 2015-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (14):
- United States (14):
  - Endocrinology Associates, Montgomery, Alabama
  - Diabetes and Endocrine Consultants P.C., Montgomery, Alabama
  - University of Miami Diabetes Research Institute, Miami, Florida
  - Dr. Rife and Associates Family Medicine, Orland Park, Illinois
  - Highland Clini-Endocrinology, Shreveport, Louisiana
  - Annapolis Internal Medicine LLC, Annapolis, Maryland
  - Nallin Family Healthcare, Cumberland, Maryland
  - Center for Diabetes and Endocrinology, Portsmouth, New Hampshire
  - North Country Community Physicians, Glen Cove, New York
  - Great Neck Medical Group, Great Neck, New York
  - North Shore Diabetes and Endocrine Associates, New Hyde Park, New York
  - Mountain Diabetes and Endocrine Center, Asheville, North Carolina
  - Primary Care Wakefield, Wakefield, Rhode Island
  - Endocrinology Associates Inc., Roanoke, Virginia